CLINICAL TRIAL: NCT03668028
Title: A Multi-center, Randomized, Independent Evaluator-Subject Blinded, Placebo-Controlled, Phase I/III Clinical Study to Evaluate Safety and Efficacy of TPX-114 for the Treatment of Full-Thickness Rotator Cuff Tear
Brief Title: A Phase I/III Clinical Study of TPX-114 for the Treatment of Full-Thickness Rotator Cuff Tear
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tego Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TPX-114-18-01; KCT0003174 (Registry Identifier: CRIS (Clinical Research Information Service, Rep. of Korea))
Record Dates: First submitted 2018-09-11; First posted 2018-09-12 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Rotator Cuff Injuries
MeSH Terms: conditions — Rotator Cuff Injuries | interventions — Arthroscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TPX-114 (Experimental): Subjects undergo arthroscopic rotator cuff repair with TPX-114.
  Interventions: Biological: TPX-114; Procedure: Arthroscopic surgery
- Placebo (Placebo Comparator): Subjects undergo arthroscopic surgery for rotator cuff repair without TPX-114.
  Interventions: Procedure: Arthroscopic surgery

INTERVENTIONS:
Biological: TPX-114 — Subjects will be treated with autologous fibroblasts (TPX-114) during arthroscopic surgery.
  Arms: TPX-114
Procedure: Arthroscopic surgery — Subjects undergo conventional arthroscopic surgery for rotator cuff repair.

SUMMARY:
Rotator cuff tear is one of the most common shoulder diseases and retears occur frequently after arthroscopic repair. Therefore, there is a growing need of new therapy to improve structural outcome. This study evaluates the efficacy and safety of autologous fibroblasts during arthroscopic repair. The primary outcome is the retear rate at 24 weeks after administration of autologous fibroblasts (TPX-114) during arthroscopic repair. Secondary outcomes are functional evaluations including Range of Motion (ROM), Constant Score (CS), American Shoulder and Elbow Surgeons (ASES) score and Simple Shoulder Test (SST) at 24 and 52 weeks after administration.

ELIGIBILITY:
Inclusion Criteria:

Participants must;

1. Be 19 years of age or older.
2. Require arthroscopic repair for full-thickness rotator cuff tear(>2cm, ≤5cm) assessed by MRI without improvement of symptoms despite more than 3 months of conservative management.
3. Consent to undergo skin biopsy to manufacture test product.
4. Understand fully the study and voluntarily sign the informed consent for participation in the study.

Exclusion Criteria:

Participants with any of the following conditions will be excluded unless stated otherwise;

1. Unsuitable for skin biopsy.
2. Have additional subscapularis tear.
3. Have prior medical history of the following at the time of screening.

   * Operation of the affected shoulder
   * Allergies to bovine proteins
   * Anaphylaxis to gentamicin
   * Coagulopathy
   * Genetic disorders affecting fibroblasts or collagen (ex. achondroplasia, osteogenesis imperfecta)
   * Malignant tumors within the last 5 years
4. Have been diagnosed with any of the following diseases at the time of screening.

   * Autoimmune disease (including RA)
   * HIV Ab-positive
   * Acute trauma, chronic shoulder dislocation, pyogenic infection on the affected shoulder
   * Scapulohumeral osteoarthritis
5. Be pregnant, breastfeeding, planning pregnancy or unwilling to use of contraceptives suggested in this study.
6. Other surgical or nonsurgical procedures on the affected shoulder to be judged more appropriate than arthroscopic repair.
7. Have participated in and received investigational agents in other clinical trials within 4 weeks of this study.
8. Be deemed inadequate for the study by investigators.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2018-07-09 (Actual); Primary Completion 2021-09-27 (Actual); Study Completion 2022-04-28 (Actual)

PRIMARY OUTCOMES:
Retear Rate | 24 weeks
  Retear rate assessed by an independent evaluator with MRI

CONTACTS AND LOCATIONS:
Overall Officials: Joo Han Oh, Principal Investigator — Seoul National University Bundang Hospital
Locations (2):
- South Korea (2):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided